CLINICAL TRIAL: NCT06761339
Title: A Randomized, Open-Label, Single-Center, Controlled Clinical Trial to Evaluate the Cough-Relieving and Expectorant Effects of the Health Supplement AZKA Nasal and Throat for Children With Outpatient-Treated Pharyngitis at Hai Phong University of Medicine and Pharmacy Hospital
Brief Title: Clinical Trial Evaluate the Cough-relieving and Expectorant Effects of the Health Supplement AZKA Nasal and Throat for Children in Outpatient-treated Pharyngitis
Acronym: AZKA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Haiphong University of Medicine and Pharmacy (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: HPMU.CTBE/P0224; 01/2024/HD/AV-YDHP (Other Grant/Funding Number: Anvy Joint Stock Company)
Record Dates: First submitted 2024-12-22; First posted 2025-01-07 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-04

CONDITIONS: Cough Severity; Cough Frequency; Cough Duration; Phlegm Accumulation (Nasal and Throat Mucus)
Keywords: Azka Nasal and Throat; Cough Relief
MeSH Terms: conditions — Cough

STUDY DESIGN:
Intervention Model Description: This clinical trial compares Azka Nasal and Throat for Children with the control drug Prospan Cough Syrup. The study duration for each participant is 15 days, which includes a 1-day screening phase, a 7-day treatment phase, and a 7-day follow-up phase after the final dose. Participants take the study products orally, 7.5 ml per dose, three times a day, 30 minutes before meals.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm 1: Azka Nasal and Throat for Children (Experimental): This arm includes 12 patients who receive the health supplement Azka Nasal and Throat for Children. Participants take the product orally, 7.5 ml per dose, three times a day, 30 minutes before meals, for 7 days.
  Interventions: Dietary Supplement: Azka Nasal and Throat for Children
- Arm 2: Prospan Cough Syrup (Active Comparator): This arm includes 12 patients who receive the control drug Prospan Cough Syrup. Participants take the product orally, 2.5 ml per dose, three times a day, 30 minutes before meals, for 7 days.
  Interventions: Drug: Prospan cough Syrup

INTERVENTIONS:
Dietary Supplement: Azka Nasal and Throat for Children — Azka Nasal and Throat for Children is provided as a liquid oral preparation, designed with a pleasant flavor to ensure compliance in pediatric patients. The intervention involves administering 7.5 ml per dose three times daily, taken orally 30 minutes before meals, for a duration of 7 days. The supplement is intended to alleviate symptoms of nasal and throat irritation, reduce phlegm, and improve overall respiratory comfort. Azka Nasal and Throat for Children has been widely used in clinical and community settings, with a favorable safety profile and reported effectiveness in pediatric respiratory care.
  Arms: Arm 1: Azka Nasal and Throat for Children
Drug: Prospan cough Syrup — The active comparator, Prospan Cough Syrup is a plant-based herbal medicinal product containing the active ingredient Hedera helix (ivy leaf extract), standardized to ensure consistent pharmacological efficacy. The syrup is formulated as an oral liquid preparation with a pleasant taste suitable for pediatric and adult use. The intervention involves administering 2.5 ml per dose three times daily, taken orally 30 minutes before meals, for a duration of 7 days.
  Arms: Arm 2: Prospan Cough Syrup

SUMMARY:
This is a randomized, open-label, single-center clinical trial evaluating the efficacy and safety of Azka Nasal and Throat for Children compared to the control drug Prospan Cough Syrup in children aged 4-6 years diagnosed with acute nasopharyngitis. Participants will be randomly assigned in a 1:1 ratio to receive either Azka Nasal and Throat or Prospan Cough Syrup for 7 days. The study aims to assess improvements in cough and phlegm conditions, as well as monitor adverse events associated with the interventions. Data will be collected over a 15-day period, including screening, treatment, and follow-up phases.

DETAILED DESCRIPTION:
This clinical trial aims to compare the efficacy and safety of Azka Nasal and Throat for Children, a registered health supplement, with Prospan Cough Syrup, a commonly used control drug. The study targets children aged 4-6 years diagnosed with acute nasopharyngitis, presenting symptoms such as cough, nasal mucus, and throat phlegm.

Participants will be randomly assigned in a 1:1 ratio to one of two arms:

Azka Nasal and Throat for Children: Administered orally at 7.5 ml per dose, three times daily, 30 minutes before meals, for 7 days.

Prospan Cough Syrup: Administered orally at 2.5 ml per dose, three times daily, 30 minutes before meals, for 7 days.

The study spans 15 days for each participant, consisting of three phases:

Screening Phase (1 day): Eligibility determined based on inclusion and exclusion criteria.

Treatment Phase (7 days): Daily administration of the assigned intervention. Follow-Up Phase (7 days): Monitoring of post-treatment outcomes. Primary outcomes include changes in cough and phlegm conditions assessed on Days 4 and 8, using the PCC scale, cough frequency, and duration of each episode, as well as the assessment of nasal and throat mucus. Secondary outcomes include the evaluation of adverse events for both interventions.

Data will be analyzed using SPSS Statistics 23.0 software to determine efficacy and safety. Descriptive statistics, t-tests, and Mann-Whitney tests will be applied based on data distribution. A significance level of p < 0.05 will be used.

This study seeks to provide valuable insights into the effectiveness of Azka Nasal and Throat for Children in improving respiratory symptoms and its safety profile compared to an established control drug.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 4-6 years. Parents or guardians agree to participate and are capable of attending study visits and assisting their children with procedures outlined in the study protocol. Parents or guardians must also agree to sign the Informed Consent Form (ICF).

A confirmed diagnosis of acute nasopharyngitis at the initial visit. Presence of symptoms such as cough, nasal mucus, and throat phlegm at the initial visit.

Exclusion Criteria:

* Complicated pharyngitis. History of malignancies in any organ system or unstable conditions that may pose risks to the participant during the study.

After screening, participants will be randomly assigned in a 1:1 ratio to one of the following interventions:

Azka Nasal and Throat for Children. Prospan Cough Syrup (control drug).

Additional Exclusions:

Planned hospitalization during the study period. Participation in a clinical trial within the past 14 days. Investigator's assessment that the participant is unsuitable for the study due to an inability to comply with the study procedures, restrictions, or requirements.

Ages: 4 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 24 (Actual)
Dates: Start 2024-12-23 (Actual); Primary Completion 2025-02-27 (Actual); Study Completion 2025-04-28 (Actual)

PRIMARY OUTCOMES:
Cough Condition Improvement Assessment | Day 4 and Day 8
  Description: Assessment of changes in cough severity, frequency, and duration using the Pediatric Cough Questionnaire (PCQ). The PCQ uses a scale ranging from 0 (Not at all) to 25 (Extremely severe). Higher scores indicate worse outcomes.
Phlegm Severity Improvement Assessment | Day 4 and Day 8
  Description: Assessment of phlegm condition using three categories:
  No Phlegm: Absence of nasal and throat mucus. Improved/Reduced: Reduction in phlegm quantity or severity. Completely Resolved: Complete resolution of phlegm symptoms. The assessment is based on clinical evaluation at baseline (Day 0), Day 4, and Day 8.

SECONDARY OUTCOMES:
Adverse Events Monitoring | Throughout the 15-Day Study Period
  Monitoring and recording of adverse events associated with Azka Nasal and Throat for Children and Prospan Cough Syrup throughout the study period.

CONTACTS AND LOCATIONS:
Locations (1):
- Center for Clinical Trial and Bioequivalence Study, Haiphong, Vietnam